CLINICAL TRIAL: NCT00001563
Title: EPOCH Chemotherapy Plus Rituximab for Previously Treated Patients With AIDS-Associated Lymphoma
Brief Title: EPOCH Chemotherapy +/- IL-12 for Previously Untreated and EPOCH Plus Rituximab for Previously Treated Patients With AIDS-Associated Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 970040; 97-C-0040; NCT00019253 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: AIDS Related Lymphoma; AIDS-Associated Lymphoma
Keywords: Lymphomagenesis; Molecular markers of drug resistance; Refractory, progressive, or relapsed HIV + NHL; AIDS-related NHL
MeSH Terms: conditions — Lymphoma, AIDS-Related; Lymphoma, Non-Hodgkin | interventions — Filgrastim; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): EPOCH-R every 3 weeks for up to 6 cycle
  Interventions: Biological: Filgrastim; Biological: Rituximab; Drug: EPOCH

INTERVENTIONS:
Biological: Filgrastim — Filgrastim after EPOCH-R from Day 6 for 10 days every cycle.
Biological: Rituximab — EPOCH-R every 3 weeks for up to 6 cycle
Drug: EPOCH — EPOCH-R every 3 weeks for up to 6 cycle

SUMMARY:
The prognosis of AIDS-related Non-Hodgkin's lymphoma is poor, especially in the relapsed setting. There is no standard treatment, and the few small studies that have been conducted have reported dismal outcomes. The purpose of this study is to pilot the use of EPOCH plus rituximab in previously treated AIDS-related lymphoma. Clinical endpoints of the study include toxicity and response. Progression-free and overall survival will be measured. Tumors will be evaluated for p53 mutations, p-16, bcl-2 expression, tumor proliferation, c-myc and EBV when possible.

DETAILED DESCRIPTION:
The prognosis of AIDS-related Non-Hodgkin's lymphoma is poor, especially in the relapsed setting. There is no standard treatment, and the few small studies that have been conducted have reported dismal outcomes. The purpose of this study is to pilot the use of EPOCH plus rituximab in previously treated AIDS-related lymphoma. Clinical endpoints of the study include toxicity and response. Progression-free and overall survival will be measured. Tumors will be evaluated for p53 mutations, p-16, bcl-2 expression, tumor proliferation, c-myc and EBV when possible.

ELIGIBILITY:
* INCLUSION CRITERIA:

Aggressive CD20 + NHL confirmed by Pathology, DCS.

HIV + serology.

All stages (I-IV) of disease.

NHL previously treated with up to two chemotherapy regimens and evaluable disease.

Age greater than or equal to 18 years.

Laboratory test: (Abnormalities are allowed if due to organ involvement by lymphoma).

Creatinine less than or equal to 1.7.

Bilirubin must be less than 2.0 mg/dl, or total bilirubin less than or equal to 3.7 mg/dl with direct fraction less than or equal to 0.2 mg/dl and indirect fraction of less than or equal 3.5 mg/dl in patients for whom these abnormalities are felt to be due to protease inhibitor therapy.

AST and ALT less than or equal to 3 times ULN (AST and ALT less than or equal to 6 times ULN for patients on hyperalimentation for whom these abnormalities are felt to be due to the hyperalimentation).

ANC greater than or equal 1000/mm(3).

Platelets must be greater than or equal to 75,000/mm(3) (patients with ITP platelets greater than or equal to 30,000/mm(3).

Signed informed consent and Durable Power of Attorney.

EXCLUSION CRITERIA:

Pregnancy or nursing.

History of clinical heart failure or symptomatic ischemic heart disease.

Serious underlying medical condition or infection other than HIV that would contraindicate EPOCH.

Concurrent anti-retroviral therapy during EPOCH therapy.

Primary CNS lymphoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 1997-01-08 (Actual); Primary Completion 2005-05-05 (Actual); Study Completion 2005-05-05 (Actual)

PRIMARY OUTCOMES:
Determination of safety profile and response rates | End of Study
  number and types of adverse events {AEs), as well as the number of patients who respond to the therapy {CR, PR, SD)

CONTACTS AND LOCATIONS:
Overall Officials: Wyndham H Wilson, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kaplan LD, Abrams DI, Feigal E, McGrath M, Kahn J, Neville P, Ziegler J, Volberding PA. AIDS-associated non-Hodgkin's lymphoma in San Francisco. JAMA. 1989 Feb 3;261(5):719-24. PMID 2536124
- [Background] Sparano JA, Wiernik PH, Strack M, Leaf A, Becker NH, Sarta C, Carney D, Elkind R, Shah M, Valentine ES, et al. Infusional cyclophosphamide, doxorubicin and etoposide in HIV-related non-Hodgkin's lymphoma: a follow-up report of a highly active regimen. Leuk Lymphoma. 1994 Jul;14(3-4):263-71. doi: 10.3109/10428199409049677. PMID 7950915
- [Background] Beral V, Peterman T, Berkelman R, Jaffe H. AIDS-associated non-Hodgkin lymphoma. Lancet. 1991 Apr 6;337(8745):805-9. doi: 10.1016/0140-6736(91)92513-2. PMID 1672911
- [Derived] Kurtz DM, Scherer F, Jin MC, Soo J, Craig AFM, Esfahani MS, Chabon JJ, Stehr H, Liu CL, Tibshirani R, Maeda LS, Gupta NK, Khodadoust MS, Advani RH, Levy R, Newman AM, Duhrsen U, Huttmann A, Meignan M, Casasnovas RO, Westin JR, Roschewski M, Wilson WH, Gaidano G, Rossi D, Diehn M, Alizadeh AA. Circulating Tumor DNA Measurements As Early Outcome Predictors in Diffuse Large B-Cell Lymphoma. J Clin Oncol. 2018 Oct 1;36(28):2845-2853. doi: 10.1200/JCO.2018.78.5246. Epub 2018 Aug 20. PMID 30125215
- [Derived] Dunleavy K, Little RF, Pittaluga S, Grant N, Wayne AS, Carrasquillo JA, Steinberg SM, Yarchoan R, Jaffe ES, Wilson WH. The role of tumor histogenesis, FDG-PET, and short-course EPOCH with dose-dense rituximab (SC-EPOCH-RR) in HIV-associated diffuse large B-cell lymphoma. Blood. 2010 Apr 15;115(15):3017-24. doi: 10.1182/blood-2009-11-253039. Epub 2010 Feb 3. PMID 20130244
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1997-C-0040.html